CLINICAL TRIAL: NCT02880748
Title: Effect of Water Exchange Method on Adenoma Miss Rates in Patients Undergoing Selective Polypectomy: a Single-centered, Randomized Controlled Study
Brief Title: Effect of Water Exchange Method on Adenoma Miss Rates in Patients Undergoing Selective Polypectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Associated professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY20162059-2
Record Dates: First submitted 2016-08-19; First posted 2016-08-26 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Adenoma
Keywords: Water exchange colonoscopy; Adenoma miss rate; Polyps
MeSH Terms: conditions — Adenoma; Polyps | interventions — Methods

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Water exchange (WE) method (Experimental): Water exchange (WE) method was used for insertion to the cecum.
  Interventions: Other: Water exchange (WE) method
- Air insufflation (AI) method (Active Comparator): Air insufflation (AI) method was used for insertion to the cecum.
  Interventions: Other: Air insufflation (AI) method.

INTERVENTIONS:
Other: Water exchange (WE) method — Water exchange (WE) method was used for insertion to the cecum. And air was insufflated to distend the lumen for inspection and biopsy or polypectomy during withdrawal procedure.
  Arms: Water exchange (WE) method
Other: Air insufflation (AI) method. — Air insufflation (AI) method was used for insertion to the cecum. And air was insufflated to distend the lumen for inspection and biopsy or polypectomy during withdrawal procedure.
  Arms: Air insufflation (AI) method

SUMMARY:
Patients with colorectal adenomas are suggested to receive polypectomy. A substantial number of adenomas may be missed in patients with polyps found by previous colonoscopy. And water exchange (WE) method may increase the detection of missed adenoma compared with traditional air insufflation (AI) colonoscopy. The investigators aim to investigate whether water exchange colonoscopy method, compared with air insufflation method, can improve the detection of missed adenomas in patients undergoing selective polypectomy.

DETAILED DESCRIPTION:
For WE method, the air pump was turned off for the full duration of insertion to avoid inadvertent air insufflations and colon elongation. Residual air in the lumen was suctioned to minimize angulations at flexures. Water at 37°C was infused with a pump (Olympus) through the biopsy channel to confirm correct tip orientation for scope advancement. The infused water was removed predominantly by suction when the colonoscope was smoothly advanced during the insertion phase, and turbid luminal water due to residual feces was exchanged by clean water until the lumen was clearly visualized. Occasionally, if it was difficult to determine whether the colonoscope tip was in the cecum, air was allowed to be insufflated for observation. If the position of the scope tip was confirmed to be not in the cecum, insufflated air would be removed by suction and the WE method would be continuously used until successful intubation.

For the AI method, water was not used, and air was insufflated during insertion.

Air was insufflated to distend the lumen for inspection and biopsy or polypectomy during withdrawal for both methods. Polyps will be removed by forceps biopsy (polyps size <3mm), cold snare technique (3-6mm) or endoscopic mucosal resection (size≥6mm).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 patients undergoing selective polypectomy

Exclusion Criteria:

* Polyps found more than 6 months
* Patients with polyposis syndrome or hereditary nonpolyposis colorectal cancer
* Patients with history of inflammatory bowel disease
* Patients with planning to undergo Endoscopic Submucosal Dissection(ESD)
* Patients not undergoing standard bowel preparation
* Patients with solid feces in the last stool after bowel preparation
* Patients considered to be high risk for bleeding during Endoscopic mucosal resection (EMR), e.g. using antiplatelet drugs (clopidogrel) within 5 days before the current colonoscopy
* Hemodynamically unstable
* Pregnant women
* Unable to provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Adenoma miss rate | 12 months
  Adenoma miss rate was calculated as the number of patients with one and more additional adenomas during polypectomy procedure divided by the total number of patients in each group.

SECONDARY OUTCOMES:
adenoma-level miss rate | 12 months
  Adenoma-level miss rate was calculated as the number of additional adenomas detected in polypectomy procedure divided by the total number of adenomas in each group.
Advanced adenoma miss rate/Miss advanced adenoma per colonoscopy | 12 months
  Advanced adenoma: any with 3 or more adenomas of any size, 1 or more large adenomas 1 cm, or 1 or more adenomas with villous architecture or highgrade dysplasia.
Adenoma per positive patient (APP) | 12 months
  The mean number of adenoma per positive patient
Quality of Bowel Preparation | 12 months
  The Boston Bowel Preparation Scale (BBPS): cleanliness of each part of the colon: 0=unprepared colon segment with mucosa not seen because of solid stool that cannot be cleared; 1=portion of mucosa of the colon segment seen, but other areas of the colon segment not well seen because of staining, residual stool, and/or opaque liquid; 2=minor amount of residual staining, small fragments of stool and/or opaque liquid, but mucosa of colon segment seen well; 3=entire mucosa of colon segment seen well with no residual staining, small fragments of stool, or opaque liquid.
Complication rate | 12 months
  Bleeding, perforation and others
Pain Scores on the Visual Analog Scale compared with previous colonoscopy | 12 months
  0 = no pain, to 10 = most severe pain

CONTACTS AND LOCATIONS:
Overall Officials: Yanglin Pan, MD, Principal Investigator — Xijing Hospital of Digestive Diseases
Locations (1):
- Endoscopic center, Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Veitch AM, Vanbiervliet G, Gershlick AH, Boustiere C, Baglin TP, Smith LA, Radaelli F, Knight E, Gralnek IM, Hassan C, Dumonceau JM. Endoscopy in patients on antiplatelet or anticoagulant therapy, including direct oral anticoagulants: British Society of Gastroenterology (BSG) and European Society of Gastrointestinal Endoscopy (ESGE) guidelines. Gut. 2016 Mar;65(3):374-89. doi: 10.1136/gutjnl-2015-311110. PMID 26873868
- [Background] Hewett DG, Rex DK. Cap-fitted colonoscopy: a randomized, tandem colonoscopy study of adenoma miss rates. Gastrointest Endosc. 2010 Oct;72(4):775-81. doi: 10.1016/j.gie.2010.04.030. Epub 2010 Jun 25. PMID 20579648
- [Derived] Ren G, Wang X, Luo H, Yao S, Liang S, Zhang L, Dong T, Chen L, Tao Q, Guo X, Han Y, Pan Y. Effect of water exchange method on adenoma miss rate of patients undergoing selective polypectomy: A randomized controlled trial. Dig Liver Dis. 2021 May;53(5):625-630. doi: 10.1016/j.dld.2020.11.012. Epub 2020 Dec 31. PMID 33390353